CLINICAL TRIAL: NCT00003478
Title: Phase I Study of Intra-Tumoral, Radiolabeled, Anti-Tenascin Monoclonal Antibody 81C6 in the Treatment of Patients With Malignant Primary Brain Tumors
Brief Title: Radiolabeled Monoclonal Antibody Therapy in Treating Patients With Primary Brain Tumors
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Purpose: Treatment
Other Study IDs: 1529; DUMC-1529-01-8R4; DUMC-1363-97-9; DUMC-1409-98-9R1; DUMC-1529-00-8R3; DUMC-1630-99-9R2; DUMC-97112; NCI-5950NS20023; NCI-G98-1471; CDR0000066515 (Other: NCI)
Record Dates: First submitted 1999-11-01; First posted 2003-01-27 (Estimated); Last update posted 2013-02-20 (Estimated); Status verified 2013-02

CONDITIONS: Brain and Central Nervous System Tumors
Keywords: recurrent adult brain tumor; adult brain stem glioma; adult medulloblastoma; adult glioblastoma; adult anaplastic astrocytoma; adult anaplastic ependymoma; adult anaplastic oligodendroglioma; adult mixed glioma; adult ependymoblastoma; adult giant cell glioblastoma; adult gliosarcoma
MeSH Terms: conditions — Central Nervous System Neoplasms; Brain Neoplasms; Medulloblastoma; Glioblastoma; Astrocytoma; Ependymoma; Oligodendroglioma; Glioma; Neuroectodermal Tumors, Primitive; Gliosarcoma | interventions — Radiotherapy

INTERVENTIONS:
Procedure: conventional surgery
Radiation: iodine I 131 monoclonal antibody 81C6
Radiation: radiation therapy

SUMMARY:
RATIONALE: Monoclonal antibodies can locate tumor cells and deliver radioactive tumor-killing substances such as radioactive iodine to them without harming normal cells.

PURPOSE: This randomized phase I/II trial is studying the side effects, best way to give, and best dose of radiolabeled monoclonal antibody and to see how well it works in treating patients with primary brain tumors.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine which one of two delivery techniques (bolus injection versus microinfusion) provides the greater distribution volume of iodine I 131 antitenascin monoclonal antibody 81C6 (I 131 MAb 81C6) administered intratumorally in patients with newly diagnosed or recurrent malignant primary brain tumors.
* Determine the maximum tolerated dose of I 131 MAb 81C6 delivered intratumorally in these patients.
* Evaluate the efficacy of I 131 MAB 81C6 delivered intratumorally in these patients.

OUTLINE: This is a randomized, dose-escalation study.

Patients are randomized to receive iodine I 131 antitenascin monoclonal antibody 81C6 (I 131 MAb 81C6) by one of two delivery techniques first, then crossover to receive the antibody by the other technique 3 days later. Each patient then receives a therapeutic dose by the most efficient method. Both methods are delivered via a stereotactically-placed intralesional catheter.

* Arm I: Bolus injection method
* Arm II: Microinfusion delivery method Cohorts of 3-6 patients receive escalating doses of I 131 MAb 81C6, with dose escalation occurring separately for each arm. After 10 patients are enrolled and the best method of administration is determined, all subsequent patients receive I 131 MAb 81C6 by that method, and the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose at which no more the 2 of 6 patients experience dose-limiting toxicity.

Patients with newly diagnosed tumors for which no effective conventional therapy exists, such as malignant glial tumors, are treated with external beam radiotherapy within 4 months after I 131 MAb 81C6 infusion. Patients with recurrent tumors receive no other therapy unless tumor progresses.

Patients are followed at 4, 8, 16, and 24 weeks and then every 12 weeks for one year.

PROJECTED ACCRUAL: At least 10 patients will be accrued for this study within 1 year.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically proven newly diagnosed or recurrent primary intracranial WHO grade III or IV glioma
* Reactivity of tumor cells with 81C6 demonstrated by immunohistology with either a polyclonal rabbit antibody or the monoclonal mouse antibody
* Radiographic evidence of a single lesion by MRI or CT scan

  * No greater than 2 to 5 cm
* No cerebral herniation syndrome
* Midline brain shift less than 0.5 cm

PATIENT CHARACTERISTICS:

Age:

* 18 and over

Performance status:

* Karnofsky 60-100%

Life expectancy:

* Not specified

Hematopoietic:

* Absolute neutrophil count greater than 1000/mm^3
* Platelet count greater than 100,000/mm^3
* Hemoglobin greater than 10 g/dL

Hepatic:

* Bilirubin less than 1.5 mg/dL
* Alkaline phosphatase less than 1.5 times normal
* SGOT less than 1.5 times normal

Renal:

* Creatinine less than 2.0 mg/dL

Other:

* Not pregnant or nursing
* Fertile patients must use effective contraception
* No allergies to iodine or local anesthetics

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* No concurrent autologous bone marrow transplant

Chemotherapy:

* No more than 1 prior conventional or phase II chemotherapy regimen
* No prior phase I chemotherapy regimens
* At least 4 weeks since prior chemotherapy
* No concurrent systemic chemotherapy

Endocrine therapy:

* Corticosteroids allowed but must be on stable dose for at least 1 week

Radiotherapy:

* At least 3 months since radiotherapy to site of measurable disease in the nervous system, unless evidence of progression

Surgery:

* Not specified

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 1997-10; Primary Completion 2007-07 (Actual); Study Completion 2007-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Darell D. Bigner, MD, PhD, Study Chair — Duke Cancer Institute
Locations (1):
- Duke Comprehensive Cancer Center, Durham, North Carolina, United States